CLINICAL TRIAL: NCT02098863
Title: Sickle Cell Clinical Research and Intervention Program
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Memphis School of Public Health (Unknown); Le Bonheur Children's Hospital (Other); University of Alabama at Birmingham (Other); Washington University School of Medicine (Other); UTHSC-ORNL Center in Biomedical Informatics (Unknown); University of Washington (Other); Medical College of Wisconsin (Other); University of Tennessee (Other); Children's Hospital of Philadelphia (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Vanderbilt University School of Medicine (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: SCCRIP; 1U01HL133996 (NIH); UTHSC-MRC Sub (Other Grant/Funding Number: Tennessee State)
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Anemia; Sickle Cell Disease; Survival; Mortality; End-Order Dysfunction
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 99 Years
Biospecimen Retention: Samples With DNA — All participants will be offered the option of having biological specimens collected and saved for future research. DNA, plasma, and urine will be collected from participants and stored in St. Jude Biorepository. In addition, buccal, nasal, and rectal swabs and stool samples will be collected from participants and stored in the Infectious Disease repository at St. Jude Children's Research Hospital. This will facilitate future high quality genotype-phenotype studies and other genetic and proteomic studies related to variability in disease severity, treatment response, and health outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the important work of previous sickle cell disease (SCD) cohort studies, there remain many understudied areas that require investigation. An important knowledge deficit is the slow but progressive process of chronic end-organ dysfunction. The majority of organ dysfunction becomes apparent in the young adult years, but comprehensive assessment of adults and understanding of predictors of adulthood organ dysfunction are insufficient. Similarly, the role of disease-modifying therapies, such as hydroxyurea, in preventing organ dysfunction later in life is not clear. Extended follow-up of patients through the transition into adulthood is imperative to understand the long-term implications of pediatric sickle cell care.

This observational study will collect data in a systematic fashion at participants' regular clinic visits (in-person or remote) to answer the objectives described below.

In addition to primary study objectives, SCCRIP participants will be eligible to participate in a sub-study, which will investigate genetically determined responses to Hydroxyurea (HU) via a pharmacokinetic study (PK). This one time study will involve blood collection at timed intervals proceeding a dose of HU. Defining the basis for this inter-individual variability will allow the identification of poor HU responders prior to initiation of therapy and the seeking of alternative treatments which seek to optimize disease treatment by accounting for individual variability in genes, environment, and lifestyle.

DETAILED DESCRIPTION:
The St. Jude Pediatric SCD Program has developed a comprehensive plan of care that spans the ages of 0 to 25, and provides the structure for screening and monitoring disease progression and complications in infancy, childhood, and young adulthood. From age 0 to 18, SCD patients are followed at St. Jude Children's Research Hospital. At age 18, their care is typically transferred to either the Methodist Adult Comprehensive Sickle Cell Disease Center in Memphis, TN, or the Regional One Health, Diggs-Kraus Sickle Cell Center in Memphis, TN, where they are routinely followed from age 18 to 25 years. After age 25, participants will be followed and invited to return to St. Jude every 6 years for study related tests until participants elect to come off study or until death.

St. Jude Children's Research Hospital, the Methodist Adult Comprehensive Sickle Cell Disease Center and the Regional One Health Diggs-Kraus Sickle Cell Center, in Memphis, TN serve as enrolling centers for the SCCRIP protocol. Two St. Jude Affiliate locations will also be sites of enrollment for this protocol for patients age 0 to 18 years. These include St. Jude Affiliate sites located in: Peoria, Illinois and Charlotte, North Carolina. Approximately 300 additional participants are expected to be enrolled from these affiliate sites. This protocol will collect data on SCD participants from birth to end of life.

The SCD plan of care provides the specific sequence of laboratory and imaging studies that are performed according to the patient's age and expected course of illness. The following health outcomes are systematically monitored in patients with SCD: hematologic indices, pulmonary function, cardiac function, renal function, cognitive function, cerebral vasculopathy, vitamin D deficiency and bone health, parvovirus B19 immune status, ophthalmologic status, and splenic function. These tests are used to direct the patient's clinical management and initiate therapies when necessary.

Participants will be administered a developmental evaluation at approximately 1 year of age. The evaluation will utilize standardized performance-based measures as well as parent rating scales lasting approximately 2 hours. Domains assessed will include cognitive, motor, language, and adaptive development.

A Neuropsychological Screener may be completed with participants within the Young Adult and Adult cohorts, every 6 years. The screening will include a series of verbal and nonverbal problem-solving activities, pencil & paper tasks, and will include a computerized component.

Quality of Life evaluations (Pediatric Quality of Life Inventory (PedsQL™) will be offered.

In this study, the results of these tests will be collected and entered into the study database, providing longitudinal data that will inform health outcomes research regarding SCD and how the course is altered by disease-modifying therapy, in addition to facilitating future interventional projects.

Primary Objectives:

* To establish a longitudinal clinical cohort of patients with sickle cell disease (SCD) to serve as a research resource to facilitate evaluation of health outcomes in SCD from pediatric care into adulthood.
* To facilitate the collection of biological samples from patients with SCD to be used in future studies investigating genetic and epigenetic contributions to disease severity, response to treatment, and morbidity and mortality.

Secondary Objectives:

* To determine the incidence, prevalence, and severity of SCD complications and adverse health conditions within the SCD cohort during five stages of development and adulthood: the newborn period (birth to 5.9 months), the infant/pre-school stage (ages 6 months to 5.9 years), the early school stage (ages 6 to 11.9 years), the adolescent stage (ages 12 to 17.9 years), young adulthood (ages 18 to 24.9 years) and mature adulthood (ages 25 and above).
* To identify and evaluate risk factors for premature mortality and long-term morbidity in patients with SCD, including those related to disease-modifying therapies, end-organ damage, genetics, neurocognitive deficits, psychosocial factors, and behavioral causes.
* To investigate the long-term effects of hydroxyurea and other therapies on preservation of organ function, growth and development, and frequency and severity of disease complications, and their long-term medical, neurocognitive, and psychosocial toxicities.
* To determine the functional aspects of the Transition to Adult Care Program within a clinical research cohort by evaluating disease specific health literacy and readiness in relation to healthcare utilization during adult care.
* To explore the long-term alterations of prolonged antibiotic exposure on the microbial community composition among people living with SCD through the collection of swabs as guided by the Human Microbiome Project (HMP) Manual of Procedures.

Other Pre-Specified Objective:

* Define the drug-exposure to clinical response relationship of HU therapy in children with SCD.

ELIGIBILITY:
SCCRIP Inclusion Criteria:

* A diagnosis of sickle cell disease of any genotype.
* PK Sub-study Inclusion Criteria:

  * Participants at St. Jude Children's Research Hospital who are consented to the parent protocol (SCCRIP, Amendment 6.1 or above).
  * Participants currently completing a hydroxyurea (HU) regimen, who have achieved maximum tolerated dose and have maintained that dose for a minimum of 90 days prior to enrollment.

SCCRIP Exclusion Criteria:

* Any medical or social reason, which, in the opinion of the principal investigators would make the participation of the subject ill-advised.
* PK Sub-study Exclusion Criteria:

  * Participants unable to complete the blood draws required for PK sampling.
  * Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
  * Any medical or social reason, which, in the opinion of the principal investigators would make the participation of the subject ill-advised.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with a diagnosis of sickle cell disease of any genotype.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-04-15 (Actual); Primary Completion 2044-12 (Estimated); Study Completion 2044-12 (Estimated)

PRIMARY OUTCOMES:
Relationship between treatment plan and health outcomes in participants with sickle cell disease (SCD) | Every 2 years from newborn to ≤ 30 years of age, and every 6 years after age 30 until end-of-life, up until December 2044
  As described in the Detailed Description, standard of care data will be collected from participants every two years during participants' annual clinic visits until study participation is discontinued or until participants reach death/end of life, whichever occurs last. This collection of observational data will be entered into a study database and will serve as a research resource to facilitate evaluation of health outcomes in participants with SCD from pediatric care into adulthood.
Relationship between genetic properties of biological samples and health outcomes in participants with sickle cell disease | Collected every 6 years from newborn until end-of life, up until December 2044
  A repository of biological samples from participants with sickle cell disease will be established for future retrospective studies investigating genetic and epigenetic contributions to disease severity, response to treatment, and morbidity and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Takemoto, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (6):
- United States (6):
  - Children's Hospital of Illinois at OSF-Saint Francis Medical Center, Peoria, Illinois
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Novant Health Hemby Children's Hospital, Charlotte, North Carolina
  - Regional One Health, Diggs-Kraus Sickle Cell Center, Memphis, Tennessee
  - Methodist Adult Comprehensive Sickle Cell Center, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Derived] Zahr RS, Kang G, Zhang X, Rashkin SR, Kovesdy CP, Takemoto C, Weiss M, Lebensburger J, Ataga KI, Saraf SL. Development of Polygenic Risk Score for Persistent Albuminuria in Children and Adults With Sickle Cell Anemia. Am J Hematol. 2025 Jun;100(6):1019-1028. doi: 10.1002/ajh.27678. Epub 2025 Apr 5. PMID 40186439
- [Derived] Chang TC, Yu J, Wang Z, Hankins JS, Weiss MJ, Wu G, Westhoff CM, Chou ST, Zheng Y. Machine learning to optimize automated RH genotyping using whole-exome sequencing data. Blood Adv. 2024 Jun 11;8(11):2651-2659. doi: 10.1182/bloodadvances.2023011660. PMID 38522094
- [Derived] Rai P, Okhomina VI, Kang G, Martinez HR, Hankins JS, Joshi V. Longitudinal effect of disease-modifying therapy on left ventricular diastolic function in children with sickle cell anemia. Am J Hematol. 2023 Jun;98(6):838-847. doi: 10.1002/ajh.26911. Epub 2023 Mar 20. PMID 36890729
- [Derived] Champlin G, Hwang SN, Heitzer A, Ding J, Jacola L, Estepp JH, Wang W, Ataga KI, Owens CL, Newman J, King AA, Davis R, Kang G, Hankins JS. Progression of central nervous system disease from pediatric to young adulthood in sickle cell anemia. Exp Biol Med (Maywood). 2021 Dec;246(23):2473-2479. doi: 10.1177/15353702211035778. Epub 2021 Aug 18. PMID 34407676
- See also: St. Jude Children's Research Hospital — http://stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols
- See also: SCCRIP: Sickle Cell Research and Intervention Program — https://www.stjude.org/research/clinical-trials/sccrip-hematological-disorder.html